CLINICAL TRIAL: NCT00352014
Title: Do Point-of-care Platelet Function Assays Predict Clinical Outcomes in Clopidogrel Pre-treated Patients Undergoing Elective PCI. (The POPular Study)
Brief Title: Evaluation and Comparison of Several Point-of-care Platelet Function Tests in Predicting Clinical Outcomes in Clopidogrel Pre-treated Patients Undergoing Elective PCI.
Status: Completed | Type: Observational
Sponsor: R&D Cardiologie (Other)
Other Study IDs: Z-05.13
Record Dates: First submitted 2006-07-13; First posted 2006-07-14 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Stable Angina Pectoris
Keywords: Monitoring of antiplatelet therapy; antiplatelet therapy; platelet function assays; Aspirin; Clopidogrel; elective PCI
MeSH Terms: conditions — Angina, Stable

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to investigate whether the level of Platelet Inhibition as assessed with five point-of-care platelet function assays correlates with clinical (periprocedural) outcomes such as Acute Myocardial Infarction, death, Target Vessel revascularization and/or stroke in patients undergoing elective PCI.

DETAILED DESCRIPTION:
Antiplatelet agents-aspirin, thienopyridines, and platelet glycoprotein IIb/IIIa (GpIIb/IIIa) inhibitors-have become cornerstones in the treatment of ischemic heart disease for patients undergoing percutaneous coronary intervention (PCI)1,2. However, several studies have demonstrated with the use of platelet function assays that subgroups of patients receiving either aspirin, clopidogrel, or both fail to produce the anticipated antiplatelet effect3-5. Consequently, terms like "aspirin-resistance" and "clopidogrel resistance" have been introduced in literature.

Light transmittance platelet aggregometry is generally considered to be the gold standard for determining platelet function, but its relevance to in vivo platelet function is questionable and the logistically demands of the method make it impossible to use in daily practice. In addition, aggregation is just one of several important platelet functions. The introduction of several point-of-care assays may be the key to the widespread clinical use of platelet function testing to identify so called anti-platelet therapy low-responders. However, whether these point-of-care platelet function tests provide predictive value (i.e. correlate with clinical outcomes) and the allocation of the "best" or most suitable point-of-care Platelet function assay to determine the level of inhibition of platelet function remains to be established.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery disease with objective evidence of ischemia (e.g., symptoms of angina pectoris, positive results of a stress test or dynamic electrocardiographic [ECG] changes)
* Adequate Aspirin and Clopidogrel pre-treatment.( Adequate clopidogrel pre-treatment is defined as a 600 mg loading dose of clopidogrel at least 6 hours prior to the PCI-procedure or a 300 mg loading dose of clopidogrel >24 hours prior to the PCI-procedure or a 75 mg dose of clopidogrel for at least >5 days prior to the PCI procedure
* Patient is thought to be at a high likelihood for requiring PCI (significant angiographic lesions in native coronary arteries amenable to and requiring a percutaneous coronary intervention)
* A stent (either drug-eluting or bare metal) is planned to be placed in at least one lesion.
* Written Informed consent

Exclusion Criteria:

* ST-segment elevation Acute Myocardial Infarction (ST-segment ≥0.1mV in ≥2 contiguous ECG leads persisting for at least 20 minutes) within 48 hours from symptom onset.
* Contraindications to antithrombotic/antiplatelet therapy
* Failed coronary intervention in the previous 2 weeks
* Malignancies
* Increased risk of bleeding (previous stroke in the past months, active bleeding or bleeding diathesis, recent trauma or major surgery in the last month, suspected aortic dissection, oral anticoagulation therapy with coumarin derivate within 7 days, recent use of GPIIb/IIIa inhibitors within 14 days, severe uncontrolled hypertension >180 mmHg unresponsive to therapy)
* Relevant hematologic deviations (hemoglobin <100g/L (6,2 mmol/L) or hematocrit <34%, platelet count <100 x 109 /L or platelet count > 600 x 109/L)
* Known allergy to clopidogrel
* Pregnancy (present or suspected)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2006-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jurrien M ten Berg, MD, PhD, Principal Investigator — Department of Cardiology, St. Antonius Hospital Nieuwegein, The Netherlands; Jochem W van Werkum, MD, Study Chair — Department of Research and Development in Cardiology, St. Antonius Hospital Nieuwegein, The Netherlands; Christian M Hackeng, PhD, Study Chair — Department of Clinical Chemistry, Nieuwegein, St. Antonius Hospital The Netherlands
Locations (1):
- Department of Cardiology, St. Antonius Hospital, The Netherlands, Nieuwegein, Utrecht, Netherlands

REFERENCES:
- [Derived] Bouman HJ, Harmsze AM, van Werkum JW, Breet NJ, Bergmeijer TO, Ten Cate H, Hackeng CM, Deneer VH, Ten Berg JM. Variability in on-treatment platelet reactivity explained by CYP2C19*2 genotype is modest in clopidogrel pretreated patients undergoing coronary stenting. Heart. 2011 Aug;97(15):1239-44. doi: 10.1136/hrt.2010.220509. Epub 2011 May 31. PMID 21628721
- [Derived] Breet NJ, van Werkum JW, Bouman HJ, Kelder JC, Harmsze AM, Hackeng CM, ten Berg JM. High on-treatment platelet reactivity to both aspirin and clopidogrel is associated with the highest risk of adverse events following percutaneous coronary intervention. Heart. 2011 Jun;97(12):983-90. doi: 10.1136/hrt.2010.220491. Epub 2011 Apr 8. PMID 21478385
- [Derived] Breet NJ, van Werkum JW, Bouman HJ, Kelder JC, Ruven HJ, Bal ET, Deneer VH, Harmsze AM, van der Heyden JA, Rensing BJ, Suttorp MJ, Hackeng CM, ten Berg JM. Comparison of platelet function tests in predicting clinical outcome in patients undergoing coronary stent implantation. JAMA. 2010 Feb 24;303(8):754-62. doi: 10.1001/jama.2010.181. PMID 20179285